CLINICAL TRIAL: NCT02732561
Title: The Efficacy of Cranial Electrostimulating Therapy for Depression and Anxiety
Brief Title: The Efficacy of Cranial Electrostimulating Therapy for Depression and Anxiety Among Homeless Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00036461
Record Dates: First submitted 2016-03-23; First posted 2016-04-08 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Sham Device (Sham Comparator): Sham device
  Interventions: Device: Sham device
- Intervention (Active Comparator): CES device. cranial electrotherapy stimulation device. Alpha Stim device
  Interventions: Device: Alpha Stim device

INTERVENTIONS:
Device: Alpha Stim device — cranial electrotherapy stimulation device
  Arms: Intervention
Device: Sham device — Sham device
  Arms: Sham Device

SUMMARY:
This is a trial of the use of cranial electrostimulating therapy for depression and anxiety among homeless adults.

DETAILED DESCRIPTION:
Cranial Electrostimulating (CES) Therapy is a Food and Drug Administration (FDA) approved treatment for depression and anxiety. However, there are no known studies on the use of this device with homeless adults. The objectives of this study are as follows: 1) to evaluate the acceptability and feasibility of CES as a treatment for homeless adults; and 2) to evaluate the efficacy of CES for the treatment of anxiety and depressive symptoms among homeless adults. Participants will be randomly assigned to one of two treatments: sham (n=10) or CES (n=10). Changes in anxiety and depressive symptoms will be evaluated over time.

ELIGIBILITY:
Inclusion Criteria:

* Competent (no legal guardian) males and females between the ages of 18 to 64
* Currently homeless or recent experience of homelessness, and symptoms of anxiety or depression

Exclusion Criteria:

* Younger than 18 and older than 65
* Patients who have attempted suicide with within the past twelve months or have active suicidal ideation will be excluded for possible safety concerns
* Self-reported illegal substance use in the past 30 days. Recent use of nicotine and alcohol will be allowed. However, those with current intoxication will be excluded
* History of a seizure disorder.
* Current history of autoimmune or endocrine disorder affecting the brain, unstable cardiac disease, history of skull fracture, or craniotomy
* Patients with pacemakers or internal electronic devices like deep brain stimulation and cochlear implants
* Women who are pregnant, nursing or planning to become pregnant
* Diagnosis of Schizophrenia or Schizoaffective disorder

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Kimball, MD, Principal Investigator — Wake Forest Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sham Device | Intervention
Started | 5 | 5
Completed | 3 | 4
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Device | Intervention | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptoms
Description: Hamilton Depression Rating Scale. The Hamilton Rating Scale for Depression is a multiple item questionnaire used to provide an indication of depression and as a guide to evaluate recovery (Hedlund, 1979). The questionnaire is designed for adults and is used to rate the severity of their depression by probing mood, feelings of guilt, suicide ideation, insomnia, agitation or retardation, anxiety, weight loss, and somatic symptoms. A score of 0-7 is considered to be normal. Scores of 20 or higher indicate moderate, severe, or very severe depression, and are usually required for entry into a clinical trial. Assessment time is estimated at 20 minutes (Hamilton, 1960). Higher values represent a worse outcome. The HAM-D form lists 21 items, the scoring is based on the first 17.Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2, with a total score range of 0-50.
Time Frame: 4 weeks
Population: Only includes matched pairs
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Sham Device | Intervention
Number analyzed (Participants) | 3 | 4
units on a scale | 13.00 [7 to 18] | 6.50 [6 to 9]

2. Primary Outcome: Anxiety
Description: Hamilton Anxiety Rating Scale. The Hamilton Anxiety Rating Scale (HAM-A) is a psychological questionnaire used by clinicians to rate the severity of a patient's anxiety (Hamilton, 1959; McDowell, Newell & & McDowell, 2006). The scale consists of 14 items designed to assess the severity of a patient's anxiety. Each of the 14 items contains a number of symptoms, and each group of symptoms is rated on a scale of zero to four, with four being the most severe (with a total score range of 0-56). All of these scores are used to compute an overarching score that indicates a person's anxiety severity (Vaccarino, 2008). A score of 17 or less indicates mild anxiety severity. A score from 18 to 24 indicates mild to moderate anxiety severity. Lastly, a score of 25 to 30 indicates a moderate to severe anxiety severity. Higher values represent a worse outcome.
Time Frame: 4 weeks
Population: includes only matched pairs
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Sham Device | Intervention
Number analyzed (Participants) | 3 | 4
units on a scale | 8.00 [6 to 15] | 6.00 [5 to 6]

ADVERSE EVENTS:
Time Frame: from first patient, first visit to last patient, last visit. Approximately 2 months.
Arm/Group | Sham Device | Intervention
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
Data analyses done usually only matched pairs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No